CLINICAL TRIAL: NCT04762485
Title: Humanized Chimeric Antigen Receptor T Cells Against CD7 for Refractory/Relapsed CD7+ Acute Leukemia
Brief Title: Humanized CD7 CAR T-cell Therapy for r/r CD7+ Acute Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: PersonGen BioTherapeutics (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGSDFYY 202101
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-01

CONDITIONS: T Lymphoblastic Leukemia/Lymphoma; Mixed Phenotype Acute Leukemia; Acute Myeloid Leukemia
Keywords: CD7 Positive; CAR-T
MeSH Terms: conditions — Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD38 positive relapsed or refractory acute leukemia (Experimental): Biological/Vaccine: Humanized CD7 CAR-T cells Split intravenous infusion of CD7 CAR-T cells [dose escalating infusion of (0.5- 10)x10^6 CD7 CAR-T cells/kg
  Interventions: Biological: Humanized CD7 CAR-T cells

INTERVENTIONS:
Biological: Humanized CD7 CAR-T cells — Split intravenous infusion of CD7 CAR-T cells [dose escalating infusion of (0.5-10)x10^6 CD7 CAR-T cells/kg

SUMMARY:
This is a prospective,open-label, single center and single arm phase 1/2 study to evaluate the efficacy and safety of T cells expressing humanized CD7 chimeric antigen receptors treatment for patients with refractory/relapsed CD7 positive acute leukemia.

DETAILED DESCRIPTION:
The patients will receive infusion of CAR T-cells targeting CD7 to confirm the safety and efficacy of CD7 CAR T-Cells in CD7+ relapsed or refractory acute leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed CD7 positive relapsed/refractory acute leukemia.
2. Age 12-65 years.
3. Eastern Cooperative Oncology Group (ECOG) score 0-2.
4. CD7 on leukemia is >30% positive detected with flow cytometry.
5. Patients with left ventricular ejection fraction ≥ 0.5 by echocardiography or grade I/II cardiovascular dysfunction according to the New York Heart Association Classification.
6. Patients with aspartate aminotransferase or glutamic-pyruvic transaminase > 3x upper limit of normal or bilirubin > 2.0 mg/dL.

Exclusion Criteria:

1. Patients are pregnant or lactating
2. Patients with congenital immunodeficiency.
3. Patients with central nervous system leukemia.
4. Patients with uncontrolled active infection.
5. Patients with active hepatitis B or hepatitis C infection.
6. Patients with HIV infection.
7. Patients with atrial or venous thrombosis or embolism.
8. Patients with myo-infarction or severe arrythmia in the recent 6 months.
9. Other comorbidities that investigators considered not suitable for this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 12 months
  Adverse events are evaluated with CTCAE V5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
  ORR includes CR, CRi, MLFS and PR. Complete remission (CR)#Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x 10^9/L; platelet count >100x10^9/L. CR with incomplete hematologic recovery (CRi)#All CR criteria except for residual neutropenia (<1.0x10^9/L) or thrombocytopenia (<100x10^9/L). Morphologic leukemia-free state (MLFS): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Cumulative incidence of relapse(CIR) | 2 years
  time from the date of achievement of a remission until the date of relapse.
the duration of CAR T-cells in vivo | 2 years
  the time of CAR-T cells' persistence in blood and the copies of CAR-T cells

CONTACTS AND LOCATIONS:
Overall Officials: xiaowen tang, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, (Select), China

REFERENCES:
- [Derived] Cao X, Dai H, Cui Q, Li Z, Shen W, Pan J, Shen H, Ma Q, Li M, Chen S, Chen J, Zhu X, Meng H, Yang L, Wu D, Tang X. CD7-directed CAR T-cell therapy: a potential immunotherapy strategy for relapsed/refractory acute myeloid leukemia. Exp Hematol Oncol. 2022 Sep 29;11(1):67. doi: 10.1186/s40164-022-00318-6. PMID 36175988